CLINICAL TRIAL: NCT03063320
Title: The Effect of Chronic Consumption of Popular Spices on Postprandial Vascular Function
Brief Title: The Effect of Spice Consumption on Postprandial Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PKE Spice PP
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Intervention Model Description: 3 period randomized cross over
Who Masked: Outcomes Assessor
Masking Description: Person assessing the outcome measures will be blinded to participant allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Spice (Active Comparator): The test meal (~1200kcal and 44g fat) will contain ~0.6g of spice blend
  Interventions: Other: Spice blend
- Moderate Spice (Experimental): The test meal (~1200kcal and 44g fat) will contain ~3.7g of spice blend
  Interventions: Other: Spice blend
- Culinary Spice (Experimental): The test meal (~1200kcal and 44g fat) will contain ~7.4g of spice blend
  Interventions: Other: Spice blend

INTERVENTIONS:
Other: Spice blend — Test spices include cardamom, coriander, cumin, ginger, paprika, red pepper, turmeric, cinnamon

SUMMARY:
A 3-period randomized cross-over, controlled feeding study will be conducted to determine the effect of chronic spice consumption on postprandial vascular function. Participants will consume three test diets containing different amounts of spice. Each treatment period will last for 4 weeks. After each diet period a meal test will be conducted. Participants will consume a meal with a spice content corresponding to the diet period they have just completed. Endothelial function will be measured at 2 and 4 hours after meal consumption. Blood samples will also be taken during the 4 hours after meal consumption for measurement of lipids, immune and inflammatory markers.

DETAILED DESCRIPTION:
A 3-period randomized cross-over, controlled feeding study will be conducted to determine the effect of chronic spice consumption on postprandial vascular function, lipid levels, immune and inflammatory markers. Participants will consume three test diets containing different amounts of spice. Each treatment period will last for 4 weeks. At baseline and after each diet period a postprandial test will be conducted. Flow mediated dilation (FMD) will conducted in the fasting state and a catheter will be inserted for blood sampling. Participants will consume a control test meal containing low spice at baseline and after each diet period the test meal will contain a level of spice that corresponds to the amount of spice consumed during the diet period. Blood samples will be taken at 30, 60, 120, 180 and 240 minutes after meal consumption, and FMD will be performed at 120 and 240 minutes.

ELIGIBILITY:
Inclusion Criteria:

Men and postmenopausal women Overweight or obese (25-35kg/m2) Non-smoking Waist circumference >= 94cm for men and >=80cm for women

At least one other of the following:

* LDL- cholesterol >130mg/dL
* CRP >1mg/L
* Triglycerides >=150mg/dL
* HDL <40mg/dL for men or <50mg/dL for women
* Systolic blood pressure >= 130mmHg or diastolic >= 85mmHg
* Fasting glucose >=100mg/dL

Exclusion Criteria:

* Diabetes (fasting glucose >126mg/dL)
* Hypertension (systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg)
* Prescribed anti-hypertensive or glucose lowering drugs
* Established cardiovascular disease, stroke, diabetes, liver, kidney or autoimmune disease
* Use of cholesterol/lipid lowering medication or supplementation (psyllium, fish oil, soy lecithin, phytoestrogens) and botanicals
* Pregnancy or lactation
* Weight loss of >=10% of body weight within the 6 months prior to enrolling in the study
* Vegetarianism

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Change in flow mediated dilation | Change from baseline at 2 hours and 4 hours after meal consumption
  Endothelial function measured by FMD

SECONDARY OUTCOMES:
Lipid and lipoproteins | Change from baseline during the 4 hours after meal consumption
  Total cholesterol, LDL cholesterol, HDL cholesterol, Triglycerides
Plasma Inflammatory cytokines | Change from baseline during the 4 hours after meal consumption
  Serum: IL-1β, IL-6, IL-10, IL-12p70, interferon-gamma, monocyte chemoattractant protein-1, macrophage inflammatory protein-1alpha, TNF-alpha, vascular endothelial growth factor
Inflammatory cytokines in isolated peripheral blood mononuclear cells | Change from baseline during the 4 hours after meal consumption
  TNF-alpha, IL-6,NF-κB, I-κB, MAP kinase, COX-2, iNOS from stimulated and unstimulated lipopolysaccharides in peripheral blood mononuclear cells. Activation status of macrophages.
Glucose | Change from baseline during the 4 hours after meal consumption
  Plasma glucose
Insulin | Change from baseline during the 4 hours after meal consumption
  Plasma insulin
Plasma antioxidants | Change from baseline during the 4 hours after meal consumption
  hydrophilic ORAC, lipophilic ORAC, total ORAC

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No